CLINICAL TRIAL: NCT01843062
Title: A Randomised, Double Blind Study to Compare the Complete Remission Rate Following a 5-Week Course of Selumetinib or Placebo and Single Dose Adjuvant Radioactive Iodine Therapy in Patients With Differentiated Thyroid Cancer
Brief Title: Comparing Complete Remission After Treatment With Selumetinib/Placebo in Patient With Differentiated Thyroid Cancer
Acronym: ASTRA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was terminated based on the findings of primary analysis at 18 months post-RAI treatment. Patients pending 3 year follow up had end of study phone call.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1532C00065; 2013-000423-14 (EudraCT Number)
Record Dates: First submitted 2013-03-14; First posted 2013-04-30 (Estimated); Results first posted 2019-04-22 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Differentiated Thyroid Cancer
Keywords: Selumetinib, Differentiated Thyroid Cancer , AZD6244
MeSH Terms: interventions — AZD 6244

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Selumetinib (Experimental): Selumetinib plus Radioactive Iodine Therapy
  Interventions: Drug: Selumetinib; Drug: Radioactive Iodine Therapy
- Placebo (Placebo Comparator): Placebo plus Radioactive Iodine Therapy
  Interventions: Drug: Placebo; Drug: Radioactive Iodine Therapy

INTERVENTIONS:
Drug: Selumetinib — 3 capsules of 25 mg strength orally twice a day for approximately 5 weeks treatment period
  Arms: Selumetinib
Drug: Placebo — 3 capsules ( to match Selumetinib capsules) orally twice a day for approximately 5 weeks treatment period
  Arms: Placebo
Drug: Radioactive Iodine Therapy — A single oral radioactive iodine dose of 100 mCI(3.7 GBq) 131I (+/-10% at the time of administration)to be administered 30 days after randomization. Additionaly, Thyrogen (Recombinant human TSH) will be used to stimulate iodine uptake according to the manufacturer's recommendation(0.9 mg intramuscular injection once a day for the 2 days prior to the dose of radioactive iodine)

SUMMARY:
The study is designed to evaluate the clinical efficacy, safety and tolerability of selumetinib with radioactive iodine therapy in patients with differentiated thyroid cancer.

DETAILED DESCRIPTION:
A Randomised, Double Blind Study to Compare the Complete Remission Rate Following a 5-Week Course of Selumetinib or Placebo and Single Dose Adjuvant Radioactive Iodine Therapy in Patients with Differentiated Thyroid Cancer.

ELIGIBILITY:
Inclusion Criteria:

Differentiated thyroid cancer Tumor >4 cm, or Gross extra-thyroid extension, or 1 lymph node >1 cm, or 5 or more lymph nodes of any size Previous thyroidectomy Must be able to receive radioactive iodine therapy Must be able to receive Thyroid Stimulating Hormone suppression

Exclusion criteria:

Metastaic disease Anaplastic thyroid cancer, medullary thyroid cancer or Hurthle cell carcinoma Presence of anti-Tg antibodies Previous treatment with any radiation Unresolved toxicity ≥ common terminology criteria for adverse event Grade 2

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2013-08-27 (Actual); Primary Completion 2018-05-18 (Actual); Study Completion 2019-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Ho, M.D., PHD, Principal Investigator — Memorial Sloan Kettering Cancer Centre, 1275 York Avenue, New York, NY 10065.; Tracy C Cunningham, M.D, Study Director — Melbourn Science Park, Cambridge Road, Melbourn, Hertfordshire, SG8 6HB, UK
Locations (42):
- United States (13):
  - Research Site, Birmingham, Alabama
  - Research Site, Little Rock, Arkansas
  - Research Site, Los Angeles, California
  - Research Site, Torrance, California
  - Research Site, Aurora, Colorado
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Boston, Massachusetts
  - Research Site, New York, New York
  - Research Site, Durham, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Nashville, Tennessee
- Brazil (6):
  - Research Site, Barretos
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, Rio de Janeiro
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Research Site, Odense C, Denmark
- France (6):
  - Research Site, Angers
  - Research Site, Bordeaux
  - Research Site, Caen
  - Research Site, Lyon
  - Research Site, Toulouse
  - Research Site, Villejuif
- Germany (3):
  - Research Site, Augsburg
  - Research Site, Essen
  - Research Site, Leipzig
- Italy (4):
  - Research Site, Catania
  - Research Site, Napoli
  - Research Site, Pisa
  - Research Site, Roma
- Poland (5):
  - Research Site, Gliwice
  - Research Site, Kielce
  - Research Site, Poznan
  - Research Site, Warsaw
  - Research Site, Zgierz
- Sweden (4):
  - Research Site, Gothenburg
  - Research Site, Linköping
  - Research Site, Lund
  - Research Site, Stockholm

REFERENCES:
- [Derived] Ho AL, Dedecjus M, Wirth LJ, Tuttle RM, Inabnet WB 3rd, Tennvall J, Vaisman F, Bastholt L, Gianoukakis AG, Rodien P, Paschke R, Elisei R, Viola D, So K, Carroll D, Hovey T, Thakre B, Fagin JA; ASTRA investigator group. Selumetinib Plus Adjuvant Radioactive Iodine in Patients With High-Risk Differentiated Thyroid Cancer: A Phase III, Randomized, Placebo-Controlled Trial (ASTRA). J Clin Oncol. 2022 Jun 10;40(17):1870-1878. doi: 10.1200/JCO.21.00714. Epub 2022 Feb 22. PMID 35192411
- See also: Statistical Analysis Plan-edition 4_Redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1176&filename=Final-D1532C00065-Statistical%20Analysis%20Plan-edition%204_Redaction-checked.pdf
- See also: Redacted CSP — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1176&filename=Final-d1532c00065-redacted%20CSP-checked.pdf
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1532C00065&attachmentIdentifier=49f06c23-25bc-4cde-bd5c-904895d052e2&fileName=Final-D1532C00065-Statistical_Analysis_Plan-edition_4_Redaction-checked-v1.0000.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study conducted between 27 Aug 2013 and 06 Mar 2019. 42 centres in 8 countries randomised patients in the study. A primary analysis was performed for the 18 months post-radioactive iodine (RAI) treatment period with a data cut-off of 18 May 2018. All primary and secondary outcome measures were reported at the time of the primary analysis.
Pre-assignment Details: Eligible patients with differentiated thyroid cancer at high risk of primary treatment failure were randomly assigned (ratio 2:1), to receive selumetinib in combination with adjuvant RAI therapy or placebo and adjuvant RAI therapy for a period of approximately 5 weeks.
Groups:
- Selumetinib 75 mg BD + RAI: Patients received selumetinib (75 milligrams [mg], orally twice daily [BD]), for a period of approximately 5 weeks. Selumetinib was to be started approximately 4 weeks prior to the planned day of RAI therapy administered as a single oral dose of 100 millicuries (mCi). To stimulate iodide uptake, patients received a recombinant human thyroid stimulating hormone (rhTSH) injection for each of the 2 days immediately prior to RAI therapy.
- Placebo + RAI: Patients received placebo capsules (to match selumetinib, orally BD), for a period of approximately 5 weeks. Placebo was to be started approximately 4 weeks prior to the planned day of RAI therapy administered as a single oral dose of 100 mCi. To stimulate iodide uptake, patients received a rhTSH injection for each of the 2 days immediately prior to RAI therapy.
Period: Overall Study
Arm/Group | Selumetinib 75 mg BD + RAI | Placebo + RAI
Started | 155 | 78
Intention to Treat (ITT) Analysis Set | 155 | 78
Safety Analysis Set | 154 | 77
BRAF/NRAS Mutation Positive Analysis Set (BRAF/NRAS positive = mutations in BRAF/NRAS oncogenes had been detected) | 91 | 51
Ongoing at Primary Analysis Data Cut-off | 134 | 71
Completed (Completed the end of study visit or end of study phone call) | 133 | 69
Not Completed | 22 | 9
Not completed — Protocol Violation | 1 | 0
Not completed — New treatment following progression | 2 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Incorrect randomisation | 1 | 0
Not completed — Withdrawal by Subject | 12 | 3
Not completed — Death | 1 | 2
Not completed — Lost to Follow-up | 2 | 4

BASELINE CHARACTERISTICS:
Population: The ITT analysis set included all randomised patients. Patients who were randomised but did not subsequently go on to receive selumetinib/placebo were included in the ITT analysis set.
Groups:
- Selumetinib 75 mg BD + RAI: Patients received selumetinib (75 mg, orally BD), for a period of approximately 5 weeks. Selumetinib was to be started approximately 4 weeks prior to the planned day of RAI therapy administered as a single oral dose of 100 mCi. To stimulate iodide uptake, patients received a rhTSH injection for each of the 2 days immediately prior to RAI therapy.
- Total: Total of all reporting groups
Arm/Group | Selumetinib 75 mg BD + RAI | Placebo + RAI | Total
Number analyzed (Participants) | 155 | 78 | 233
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.2 (14.20) | 47.9 (14.67) | 46.8 (14.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 40 | 132
  Male | 63 | 38 | 101
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 14 | 41
  Not Hispanic or Latino | 128 | 64 | 192
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 145 | 73 | 218
  Black or African American | 3 | 1 | 4
  Asian | 3 | 3 | 6
  Other | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission Rate (Expressed as Percentage of Patients in Complete Remission) at 18 Months Post-RAI Treatment; ITT Analysis Set
Description: Patients were defined to be in complete remission if all of the following criteria were demonstrated:
  1. Serum thyroglobulin (Tg) levels <1 nanograms / millilitre (ng/mL) during rhTSH stimulation, in the absence of interfering Tg antibodies, as assessed by standardised central laboratory analysis.
  2. No confirmed evidence of thyroid cancer on neck ultrasound, as assessed by investigator site review.
  3. No confirmed radiological evidence of thyroid cancer, as assessed by blinded independent central review.
  4. No histopathological evidence of thyroid cancer on fine needle aspiration (FNA)/biopsy when performed, as assessed by investigator site review.
  5. No further thyroid cancer therapy was administered in the first 18 months following the initial RAI treatment.
Time Frame: At 18 months post-RAI treatment
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Selumetinib 75 mg BD + RAI | Placebo + RAI
Number analyzed (Participants) | 155 | 78
Percentage of participants | 40.0 | 38.5
Statistical Analysis 1: Comparison: Selumetinib 75 mg BD + RAI vs Placebo + RAI; Selumetinib in combination with RAI was compared with placebo in combination with RAI. The analysis was performed using a logistic regression model including treatment as the only covariate. An odds ratio >1 favours selumetinib in combination with RAI; Test type: Superiority; p = 0.8205, Regression, Logistic — The primary endpoint was to be considered statistically significant if the 2-sided p-value was less than 0.05. P-value and confidence intervals (CIs) were calculated using profile likelihood; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.61 to 1.87]

2. Secondary Outcome: Complete Remission Rate (Expressed as Percentage of Patients in Complete Remission) at 18 Months Post-RAI Treatment; Subgroup Analysis BRAF/NRAS Mutation Positive
Description: Patients were defined to be in complete remission if all of the following criteria were demonstrated:
  1. Serum Tg levels <1 ng/mL during rhTSH stimulation, in the absence of interfering Tg antibodies, as assessed by standardised central laboratory analysis.
  2. No confirmed evidence of thyroid cancer on neck ultrasound, as assessed by investigator site review.
  3. No confirmed radiological evidence of thyroid cancer, as assessed by blinded independent central review.
  4. No histopathological evidence of thyroid cancer FNA/biopsy when performed, as assessed by investigator site review.
  5. No further thyroid cancer therapy was administered in the first 18 months following the initial RAI treatment.
Time Frame: At 18 months post-RAI treatment
Population: The BRAF/NRAS mutation positive analysis set included only those patients from the ITT population whose tumour samples were mutation positive for the oncogenes BRAF or NRAS.
Measure: Number; unit: Percentage of participants
Arm/Group | Selumetinib 75 mg BD + RAI | Placebo + RAI
Number analyzed (Participants) | 91 | 51
Percentage of participants | 37.4 | 41.2
Statistical Analysis 1: Comparison: Selumetinib 75 mg BD + RAI vs Placebo + RAI; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.6549, Regression, Logistic — P-value and CIs were calculated using profile likelihood; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.42 to 1.73]

3. Secondary Outcome: Clinical Remission Rate (Expressed as Percentage of Patients in Clinical Remission) at 18 Months Post-RAI Treatment; ITT Analysis Set
Description: Patients were defined to be in clinical remission if all of the following criteria were demonstrated:
  1. Serum Tg levels <1 ng/mL during rhTSH stimulation, in the absence of interfering Tg antibodies, as assessed by standardised central laboratory analysis.
  2. No confirmed evidence of thyroid cancer on neck ultrasound, as assessed by investigator site review.
  3. No evidence of thyroid cancer on diagnostic whole body scan (WBS), as assessed by blinded independent central review.
  4. No histopathological evidence of thyroid cancer on FNA/biopsy when performed to clarify equivocal ultrasound findings, as assessed by investigator site review.
  5. No further thyroid cancer therapy was administered in the first 18 months following the initial RAI treatment.
Time Frame: At 18 months post-RAI treatment
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Selumetinib 75 mg BD + RAI | Placebo + RAI
Number analyzed (Participants) | 155 | 78
Percentage of participants | 40.0 | 38.5
Statistical Analysis 1: Comparison: Selumetinib 75 mg BD + RAI vs Placebo + RAI; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.8205, Regression, Logistic — P-value and CIs were calculated using profile likelihood; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.61 to 1.87]

4. Secondary Outcome: Clinical Remission Rate (Expressed as Percentage of Patients in Clinical Remission) at 18 Months Post-RAI Treatment; Subgroup Analysis BRAF/NRAS Mutation Positive
Description: Patients were defined to be in clinical remission if all of the following criteria were demonstrated:
  1. Serum Tg levels <1 ng/mL during rhTSH stimulation, in the absence of interfering Tg antibodies, as assessed by standardised central laboratory analysis.
  2. No confirmed evidence of thyroid cancer on neck ultrasound, as assessed by investigator site review.
  3. No evidence of thyroid cancer on diagnostic WBS, as assessed by blinded independent central review.
  4. No histopathological evidence of thyroid cancer on FNA/biopsy when performed to clarify equivocal ultrasound findings, as assessed by investigator site review.
  5. No further thyroid cancer therapy was administered in the first 18 months following the initial RAI treatment.
Time Frame: At 18 months post-RAI treatment
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Selumetinib 75 mg BD + RAI | Placebo + RAI
Number analyzed (Participants) | 91 | 51
Percentage of participants | 37.4 | 41.2
Statistical Analysis 1: Comparison: Selumetinib 75 mg BD + RAI vs Placebo + RAI; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.6549, Regression, Logistic — P-value and CIs were calculated using profile likelihood; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.42 to 1.73]

ADVERSE EVENTS:
Time Frame: Includes adverse events (AEs) with an onset date on or after the date of first dose and up to and including 30 days following the date of last dose of selumetinib/placebo. Overall timeframe for collection of AEs was up to 66 days from the first dose.
Description: All-Cause Mortality is reported for the ITT analysis set for the overall study period. Serious and Other (non-serious) AE data is reported for the safety analysis set (including all patients who received at least 1 dose of randomised treatment) for the 5-week treatment period plus 30-day follow-up phase.
Arm/Group | Selumetinib 75 mg BD + RAI | Placebo + RAI
All-Cause Mortality (participants affected / at risk) | 1/155 | 2/78
Serious Adverse Events (participants affected / at risk) | 7/154 | 0/77
Other Adverse Events (participants affected / at risk) | 141/154 | 43/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selumetinib 75 mg BD + RAI (N=154) | Placebo + RAI (N=77)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selumetinib 75 mg BD + RAI (N=154) | Placebo + RAI (N=77)
Periorbital oedema (Eye disorders) | 8 (8) | 0 (0)
Constipation (Gastrointestinal disorders) | 15 (15) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 68 (78) | 12 (13)
Dry mouth (Gastrointestinal disorders) | 15 (15) | 3 (3)
Rash follicular (Skin and subcutaneous tissue disorders) | 13 (13) | 0 (0)
Dysgeusia (Nervous system disorders) | 6 (6) | 4 (4)
Rash macular (Skin and subcutaneous tissue disorders) | 12 (12) | 2 (2)
Vision blurred (Eye disorders) | 16 (16) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 8 (8) | 1 (1)
Nausea (Gastrointestinal disorders) | 44 (44) | 8 (10)
Stomatitis (Gastrointestinal disorders) | 17 (18) | 4 (4)
Vomiting (Gastrointestinal disorders) | 14 (14) | 0 (0)
Face oedema (General disorders) | 9 (9) | 0 (0)
Fatigue (General disorders) | 44 (44) | 13 (13)
Oedema peripheral (General disorders) | 30 (32) | 4 (4)
Blood creatine phosphokinase increased (Investigations) | 31 (31) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Headache (Nervous system disorders) | 8 (8) | 10 (11)
Paraesthesia (Nervous system disorders) | 4 (4) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Acne (Skin and subcutaneous tissue disorders) | 13 (13) | 2 (2)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 67 (70) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 12 (12) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 21 (21) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 19 (19) | 4 (4)
Hypertension (Vascular disorders) | 20 (23) | 3 (3)

LIMITATIONS AND CAVEATS:
The study was terminated early (based on the findings of the primary analysis at 18 months post-RAI treatment) and all randomised patients who had not yet completed their 3-year follow-up visit were instead to have an end of study phone call.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If the Study is part of a multi-centre clinical trial, the Institution or Investigator agree not to independently publish results of, or make presentations related to, the Study until first occurrence of one of the following: multi-centre primary Publication is published; no multi-centre primary Publication is submitted within 2 years after conclusion, abandonment or termination of the Study at all sites; or Sponsor confirms in writing there will be no multi-centre primary Publication.

DOCUMENTS (2):
  • Study Protocol (2013-01-24): https://cdn.clinicaltrials.gov/large-docs/62/NCT01843062/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-04): https://cdn.clinicaltrials.gov/large-docs/62/NCT01843062/SAP_001.pdf